CLINICAL TRIAL: NCT04215250
Title: Accuracy of CVC Depth Prediction in Internal Jugular Veins: The Difference Between The Andropoulos and ECG Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Anesthesiologist Consultant, Indonesia University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IndonesiaUAnes 042
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Depth of CVC Insertion
MeSH Terms: interventions — Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Andropulous method (Active Comparator): Andropulous method uses equations to determine the depth of CVC insertion.
  For subject with <100 cm in height:
  Depth of CVC insertion (cm) = (height (cm)/ 10)-1
  For subject with >100 cm in height:
  Depth of CVC insertion (cm) = (height (cm)/ 10)-2
  Interventions: Other: andropulous method
- ECG method (Active Comparator): change in p wave from ECG
  Interventions: Device: ECG

INTERVENTIONS:
Other: andropulous method — Counts the CVC depth using specific equation
  Arms: Andropulous method
Device: ECG — Using ECG to monitor the insertion of the CVC
  Arms: ECG method

SUMMARY:
compare the accuracy of CVC depth prediction in internal jugular veins: the difference between the andropoulos and ECG methods

DETAILED DESCRIPTION:
seventy two subjects were given informed consent before the study started. compare the accuracy of CVC depth prediction in internal jugular veins with two difference methods, the andropoulos method and ECG method.

ELIGIBILITY:
Inclusion Criteria:

* signing informed consent form
* indicated for CVC insertion
* has no contraindication for right internal jugular vein CVC insertion

Exclusion Criteria:

* has history of arrhythmia
* has cardiac malformation history

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
CVC prediction depth using andropulous equation | 30 minutes
  CVC will be inserted in certain depth according to the calculated depth

SECONDARY OUTCOMES:
ECG change | 30 seconds
  changes in p wave during CVC insertion

CONTACTS AND LOCATIONS:
Overall Officials: Aida R Tantri, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang L, Liu ZS, Wang CA. Malposition of Central Venous Catheter: Presentation and Management. Chin Med J (Engl). 2016 Jan 20;129(2):227-34. doi: 10.4103/0366-6999.173525. No abstract available. PMID 26830995
- [Result] Chaskar V, Karnik PP, Dave NM, Garasia M. Comparative Study of Three Methods for Depth of Central Venous Catheter Placement in Children: An Observational Pilot Study. Turk J Anaesthesiol Reanim. 2018 Apr;46(2):116-120. doi: 10.5152/TJAR.2018.32748. Epub 2018 Apr 1. PMID 29744246
- [Result] Kwon HJ, Jeong YI, Jun IG, Moon YJ, Lee YM. Evaluation of a central venous catheter tip placement for superior vena cava-subclavian central venous catheterization using a premeasured length: A retrospective study. Medicine (Baltimore). 2018 Jan;97(2):e9600. doi: 10.1097/MD.0000000000009600. PMID 29480861
- [Result] Sharma D, Singh VP, Malhotra MK, Gupta K. Optimum depth of central venous catheter - Comparision by pere's, landmark and endocavitory (atrial) ECG technique: A prospective study. Anesth Essays Res. 2013 May-Aug;7(2):216-20. doi: 10.4103/0259-1162.118966. PMID 25885836
- [Result] Na HS, Kim JT, Kim HS, Bahk JH, Kim CS, Kim SD. Practical anatomic landmarks for determining the insertion depth of central venous catheter in paediatric patients. Br J Anaesth. 2009 Jun;102(6):820-3. doi: 10.1093/bja/aep078. Epub 2009 Apr 19. PMID 19380312
- [Result] Kremser J, Kleemann F, Reinhart K, Schummer W. Optimized method for correct left-sided central venous catheter placement under electrocardiographic guidance. Br J Anaesth. 2011 Oct;107(4):567-72. doi: 10.1093/bja/aer189. Epub 2011 Jun 22. PMID 21697183
- [Result] Andropoulos DB, Bent ST, Skjonsby B, Stayer SA. The optimal length of insertion of central venous catheters for pediatric patients. Anesth Analg. 2001 Oct;93(4):883-6. doi: 10.1097/00000539-200110000-00016. PMID 11574350
- [Result] Struck MF, Schmidt T, Winkler BE, Reinhart K, Schummer W. Formulas for prediction of insertion depths of internal jugular vein catheters adjusted to body height categories. J Vasc Access. 2016 Mar-Apr;17(2):191-4. doi: 10.5301/jva.5000488. Epub 2015 Dec 7. PMID 26660038